CLINICAL TRIAL: NCT00991523
Title: Protein Ingestion Prior to Sleep as a Dietary Strategy to Improve Post-exercise, Overnight Recovery.
Brief Title: Overnight Post-Exercise Recovery After Protein Ingestion Prior to Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Luc van Loon, University Hospital Maastricht
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: MEC 09-3-054
Record Dates: First submitted 2009-10-06; First posted 2009-10-08 (Estimated); Last update posted 2011-04-20 (Estimated); Status verified 2011-04

CONDITIONS: Exercise; Resistance Training
Keywords: resistance; exercise; protein; recovery
MeSH Terms: conditions — Motor Activity | interventions — Proteins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sweetened beverage (Experimental)
  Interventions: Dietary Supplement: protein
- placebo control (Placebo Comparator): placebo
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: protein — protein
  Arms: sweetened beverage
Dietary Supplement: placebo — placebo control
  Arms: placebo control

SUMMARY:
The purpose of this study is to examine the effects of post-exercise protein ingestion prior to sleep on overnight protein kinetics and muscle recovery.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age between 20 and 30 years
* Healthy, recreationally active
* BMI <25 kg/m2

Exclusion Criteria:

* Use of medication

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-08 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
muscle protein synthesis | 10 hours

CONTACTS AND LOCATIONS:
Overall Officials: Luc van Loon, PhD, Principal Investigator — Maastricht University Medical Center
Locations (2):
- Netherlands (2):
  - Maastricht MUMC, Maastricht, LI
  - MaastrichtUMC, Maastricht

REFERENCES:
- [Derived] Gorissen SHM, Trommelen J, Kouw IWK, Holwerda AM, Pennings B, Groen BBL, Wall BT, Churchward-Venne TA, Horstman AMH, Koopman R, Burd NA, Fuchs CJ, Dirks ML, Res PT, Senden JMG, Steijns JMJM, de Groot LCPGM, Verdijk LB, van Loon LJC. Protein Type, Protein Dose, and Age Modulate Dietary Protein Digestion and Phenylalanine Absorption Kinetics and Plasma Phenylalanine Availability in Humans. J Nutr. 2020 Aug 1;150(8):2041-2050. doi: 10.1093/jn/nxaa024. PMID 32069356
- [Derived] Res PT, Groen B, Pennings B, Beelen M, Wallis GA, Gijsen AP, Senden JM, VAN Loon LJ. Protein ingestion before sleep improves postexercise overnight recovery. Med Sci Sports Exerc. 2012 Aug;44(8):1560-9. doi: 10.1249/MSS.0b013e31824cc363. PMID 22330017